CLINICAL TRIAL: NCT05990712
Title: A Prospective Study on the Effect of Pre-cataract Surgical Ocular Hygiene Regime on Microbial Load, Tear Osmolarity, Dry Eye, and Inflammatory Markers Between Two Ocular Hygiene Regimen Groups
Brief Title: The Effect of a Pre-cataract Surgical Ocular Hygiene Regime on Microbial Load, Tear Osmolarity, Dry Eye, and Inflammatory Markers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uptown Eye Specialists (Other)
Collaborators: WIlliam Osler Health Systems (Unknown); Forsee Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UptownEye4
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Dry Eye; Dry Eye Syndromes; Cataract
Keywords: Pre-operative; Ocular hygiene; Omega 3; Microbial load; Inflammation; Tear osmolarity
MeSH Terms: conditions — Dry Eye Syndromes; Cataract; Inflammation | interventions — Docosahexaenoic Acids; Trehalose

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to either the omega-3 group or no omega-3 group.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Omega-3 (Experimental): Participants in this arm will take oral omega-3 supplement for 4 weeks pre-operatively and 4 weeks post-operatively. They will also receive the Zocular intervention in clinic and the lid wipe and Thealoz eyedrops at home.
  Interventions: Dietary Supplement: Omega-3; Drug: Trehalose; Drug: Zocular Eyelid System Treatment; Other: Blephadex cleansing eyelid wipes
- No Omega-3 (Active Comparator): Participants in this arm will not take oral omega-3 supplement. They will only receive the Zocular intervention in clinic and the lid wipe and Thealoz eyedrops at home.
  Interventions: Drug: Trehalose; Drug: Zocular Eyelid System Treatment; Other: Blephadex cleansing eyelid wipes

INTERVENTIONS:
Dietary Supplement: Omega-3 — Omega-3 is a fatty acid and there is evidence that the consumption of re-esterified oral omega-3 supplements over the course of 6 to 8 weeks aid in reducing inflammation, dry eye, and optimizing tear osmolarity. The oral omega-3 supplement taken daily.
  Arms: Omega-3
Drug: Trehalose — Eyedrops consisting of trehalose and sodium hyaluronate that lubricate and hydrate the eye to relieve dry eye.
  Other Names: Thealoz Duo Drops
Drug: Zocular Eyelid System Treatment — A lid cleaning and debridement system that consists of okra-based gel to relieve dry eye or inflammation. The gel is applied to the eyelid margin and lashes with a cotton swab.
  Other Names: ZEST
Other: Blephadex cleansing eyelid wipes — Eyelid cleansing wipes with tea tree oil and coconut that help reduce infection.

SUMMARY:
This study assesses the impact of two differing ocular hygiene regimens prior to cataract surgery. The first regimen includes an omega-3 supplement and the second without, and both include an at-home lid wipe and cleansing eye drops. These regimens will be assessed on microbial load, inflammation, tear osmolarity, and dry eye metrics. Patients will be randomized to either the omega-3 group + 3-part hygiene regimen, or the group with only the 3-part hygiene regimen. Data will be collected for inflammation through a test (InflammaDry) that measures an inflammatory marker, dry eye metrics via an imaging tool called Oculus 5M and the Canadian Dry Eye Assessment (CDEA) questionnaire, tear osmolarity through Tear Labs device, and area of growth for conjunctiva microbial load by swabbing the conjunctiva of the eye. Dry eye metrics (CDEA and Oculus 5M) will be collected during the patient's baseline appointment, 2-5 days prior to surgery, and post-operative month 1. Microbial load swabs will be collected at baseline, 2-5 days prior to surgery, and date of the surgery. An ocular assessment will also be completed at baseline, one week post-operation, and one month post-operation. All metrics will be compared to the fellow eye. The usage of omega-3 will be compared to the regimen without omega-3.

DETAILED DESCRIPTION:
Prospective interventional study assessing the impact of two ocular hygiene regimens, with and without Omega-3, on microbial load, inflammation, tear osmolarity, and dry eye metrics and disease for patients soon to undergo cataract surgery. Study recruitment will occur at Uptown Eye between Sept-Nov 2023, with a target of 68 patients enrolled in the study. Patients will be consecutively randomized to group 1 (without omega 3 group) or group 2 (with omega 3 group). The intervention includes Zocular in clinic at baseline, Thealoz Duo eyedrops twice daily until surgery, and the cleansing wipes twice daily until surgery. The omega 3 group will take the supplement from baseline until one month post-operative.

Data will be collected for inflammation through a InflammaDry Matrix metallopeptidase 9 (MMP-9) test, dry eye through Oculus 5M (measures non-invasive break-up time (NIBUT), lipid layer, bulbar redness, tear meniscus height) and Canadian Dry Eye Assessment (CDEA), TearLab for osmolarity, and conjunctival swabs for microbial load. Dry eye metrics (CDEA and Oculus 5M) will be collected during the patient's baseline Cataract Dry Eye Clinic (CDEC) appointment, 2-5 days prior to surgery, and post-operative month 1. Microbial load will be collected at baseline, 2-5 days prior to surgery, and date of the surgery. Tear osmolarity and inflammation markers will be collected at baseline, 2-5 days prior to surgery, and post-operative month. An ocular assessment will also be completed at baseline, one week post-operation, and post-operative month. All metrics will be compared to the fellow eye.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 or older who underwent cataract surgical ocular hygiene treatment regimen prior to cataract surgery.
* Patients of all severity of dry eye will be included.

Exclusion Criteria:

* Patients with any other ocular comorbidities (glaucoma, iritis, traumatic eye injury, known systemic autoimmune diseases, immune disorders, anti-inflammatory medications, blood disorders (eg. altered white counts), prior surgery, prior traumatic eye injury, previous dry eye interventions such as ocular plugs, radiofrequency, and IPL).
* Patients who have any complications arise during the cataract surgery.
* Patients with altered mental state and cannot provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
MMP-9 | Baseline, 2-5 days prior to surgery, post-operative month 1
  Level of MMP-9, an inflammatory marker reported as positive (level of MMP-9 > 40ng/mL) or negative (level of MMP-9 < 40ng/mL).
Microbial load | Baseline, 2-5 days prior to surgery, surgery day
  Area of microbial growth from conjunctival swab reported as percentage of dish coverage, incubated for 48 hours
Tear osmolarity | Baseline, 2-5 days prior to surgery, surgery day
  Measure of salt concentration in tear reported as mOsm/L

SECONDARY OUTCOMES:
Non-invasive break-up time (NIBUT) | Baseline, 2-5 days prior to surgery, post-operative month 1
  Non-invasive break-up time (NIBUT) is measured using the Oculus 5M and measured in seconds, with longer NIBUT representing better outcomes.
Lipid layer | Baseline, 2-5 days prior to surgery, post-operative month 1
  Lipid layer is reported in nanometres with higher/thicker lipid layers representing a better outcome.
Bulbar redness | Baseline, 2-5 days prior to surgery, post-operative month 1
  Bulbar redness is reported by a score from 0-4 with lower scores representing a better outcome.
Tear meniscus height | Baseline, 2-5 days prior to surgery, post-operative month 1
  Tear meniscus height (TMH) is reported in millimetres, with increases in TMH representing a better outcome.
Canadian Dry Eye Assessment (CDEA) Questionnaire | Baseline, 2-5 days prior to surgery, post-operative month 1
  12 item questionnaire for reporting of dry eye symptoms on a scale of 0-4. Total scores for the CDEA questionnaire range from 0 to 48 and are interpreted as no dry eye symptoms or normal (<5), mild dry eye symptoms (5-20), moderate dry eye symptoms (21-30), or severe dry eye symptoms (31-48).

CONTACTS AND LOCATIONS:
Locations (1):
- Uptown Eye, Brampton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No